CLINICAL TRIAL: NCT01193257
Title: A Phase 3, Randomized, Double-Blind, Multicenter Trial Comparing Orteronel (TAK-700) Plus Prednisone With Placebo Plus Prednisone in Patients With Metastatic Castration-Resistant Prostate Cancer That Has Progressed During or Following Docetaxel-based Therapy.
Brief Title: Study Comparing Orteronel Plus Prednisone in Participants With Metastatic Castration-Resistant Prostate Cancer.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C21005; 2010-018662-23 (EudraCT Number); CTR20131423 (Registry Identifier: SFDA CTR); 0991413212 (Registry Identifier: TCTIN); C21005 (Registry Identifier: NRES); U1111-1181-8040 (Registry Identifier: WHO)
Record Dates: First submitted 2010-08-31; First posted 2010-09-01 (Estimated); Results first posted 2018-12-19 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-11

CONDITIONS: Prostate Cancer
Keywords: Drug therapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — orteronel; Prednisone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Orteronel + prednisone (Experimental)
  Interventions: Drug: Orteronel; Drug: Prednisone
- Placebo + prednisone (Placebo Comparator)
  Interventions: Drug: Prednisone; Drug: Orteronel Placebo

INTERVENTIONS:
Drug: Orteronel — Orteronel tablets
  Other Names: TAK-700
  Arms: Orteronel + prednisone
Drug: Prednisone — Prednisone tablets
Drug: Orteronel Placebo — Orteronel placebo-matching tablets
  Arms: Placebo + prednisone

SUMMARY:
This is a randomized, double-blind, multicenter, phase 3 study evaluating orteronel plus prednisone compared with placebo plus prednisone in men with metastatic, castration-resistant prostate cancer (mCRPC) that has progressed following Docetaxel-based therapy

ELIGIBILITY:
Inclusion Criteria:

Each participant must meet all of the following inclusion criteria:

* Voluntary written consent
* Male 18 years or older
* Histologically or cytologically confirmed diagnosis of prostate adenocarcinoma
* Radiograph-documented metastatic disease
* Progressive disease
* Prior surgical castration or concurrent use of an agent for medical castration
* Progressive disease during or following 1 or 2 regimens of cytotoxic chemotherapy, 1 of which must have included docetaxel. Must have received greater than or equal to (>=) 360 milligram per square meter (mg/m^2) of docetaxel within a 6-month period. Participants who were clearly intolerant to docetaxel or develop progressive disease before receiving >= 360 mg/m^2 are also eligible if they have received at least 225 mg/m^2 of docetaxel within a 6-month period and meet the other study entry criteria.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2
* Even if surgically sterilized, participants must practice effective barrier contraception during the entire study treatment period and for 4 months after the last dose of study drug, OR Abstain from heterosexual intercourse
* Screening laboratory values as specified in protocol
* Stable medical condition
* Life expectancy of 6 months or more
* Participants who have had up to 2 prior chemotherapy treatments are eligible to participate

Exclusion Criteria:

Participants meeting any of the following exclusion criteria are not to be enrolled in the study:

* Known hypersensitivity to orteronel, prednisone or gonadotropin-releasing hormone (GnRH) analogue
* Received prior therapy with orteronel, aminoglutethimide, ketoconazole or abiraterone
* Any other therapies for prostate cancer, except for GnRH analogue therapy, must be discontinued 2 weeks before the first dose of study drug
* Radioisotope therapy or external beam radiation therapy within 4 weeks of first dose of study drug
* Documented central nervous system metastases
* Treatment with any investigational compound within 30 days prior to first dose of study drug (Participants who are in long-term follow-up following active treatment in other trials are eligible)
* Diagnosis or treatment of another malignancy within 2 years preceding first dose of study drug except nonmelanoma skin cancer or in situ malignancy completely resected
* Uncontrolled cardiovascular condition as specified in study protocol
* Known history of human immunodeficiency virus (HIV) infection, hepatitis B, or hepatitis C
* Unwilling or unable to comply with protocol
* Known gastrointestinal disease or procedure that could interfere with oral absorption or tolerance of orteronel
* Uncontrolled nausea, vomiting, or diarrhea despite appropriate medical therapy
* Prostate cancer confined to just the prostrate bed or immediate adjacent tissue

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1099 (Actual)
Dates: Start 2010-11-15 (Actual); Primary Completion 2013-05-16 (Actual); Study Completion 2016-02-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Millennium Pharmaceuticals, Inc.
Locations (77):
- United States (36):
  - Anchorage, Alaska
  - Fort Smith, Arkansas
  - Fountain Valley, California
  - Los Angeles, California
  - Riverside, California
  - San Diego, California
  - Fort Myers, Florida
  - Port Saint Lucie, Florida
  - Indianapolis, Indiana
  - Jeffersonville, Indiana
  - New Orleans, Louisiana
  - Westminster, Maryland
  - Detroit, Michigan
  - Jefferson City, Missouri
  - Las Vegas, Nevada
  - Hackensack, New Jersey
  - Albany, New York
  - East Syracuse, New York
  - Rochester, New York
  - Raleigh, North Carolina
  - Cincinnati, Ohio
  - Tualatin, Oregon
  - Lancaster, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Greenville, South Carolina
  - Chattanooga, Tennessee
  - Nashville, Tennessee
  - Amarillo, Texas
  - Bedford, Texas
  - Dallas, Texas
  - Odessa, Texas
  - Tyler, Texas
  - Webster, Texas
  - Salt Lake City, Utah
  - Newport News, Virginia
  - Kennewick, Washington
- Australia (5):
  - Redcliffe, Queensland
  - Woodville South, South Australia
  - Hobart, Tasmania
  - Malvere, Victoria
  - Wodonga, Victoria
- Belgium (4):
  - Brussels
  - Kortijk
  - Liège
  - Namur
- Canada (8):
  - Edmonton, Alberta
  - Kelowna, British Columbia
  - Moncton, New Brunswick
  - Brampton, Ontario
  - Newmarket, Ontario
  - Greenfield Park, Quebec
  - Montreal, Quebec
  - Pointe-Claire, Quebec
- Czechia (5):
  - Hradec Dralove
  - Kromertz
  - Modřice
  - Prague
  - Zlín
- Tallinn, Estonia
- Finland (2):
  - Oulu
  - Tampere
- France (6):
  - La Roche-sur-Yon
  - Le Mans
  - Lyon
  - Marseille
  - Paris
  - Villejuif
- Pátrai, Greece
- Hungary (2):
  - Miskolc
  - Osztaly
- Italy (2):
  - Novara
  - Rome
- Eindhoven, Netherlands
- Poland (3):
  - Bielsko-Biala
  - Goczałkowice Zdrój
  - Wroclaw
- Seville, Spain

REFERENCES:
- [Derived] Heller G, McCormack R, Kheoh T, Molina A, Smith MR, Dreicer R, Saad F, de Wit R, Aftab DT, Hirmand M, Limon A, Fizazi K, Fleisher M, de Bono JS, Scher HI. Circulating Tumor Cell Number as a Response Measure of Prolonged Survival for Metastatic Castration-Resistant Prostate Cancer: A Comparison With Prostate-Specific Antigen Across Five Randomized Phase III Clinical Trials. J Clin Oncol. 2018 Feb 20;36(6):572-580. doi: 10.1200/JCO.2017.75.2998. Epub 2017 Dec 22. PMID 29272162
- [Derived] Suri A, Chapel S, Lu C, Venkatakrishnan K. Physiologically based and population PK modeling in optimizing drug development: A predict-learn-confirm analysis. Clin Pharmacol Ther. 2015 Sep;98(3):336-44. doi: 10.1002/cpt.155. Epub 2015 Jul 14. PMID 26031410
- [Derived] Fizazi K, Jones R, Oudard S, Efstathiou E, Saad F, de Wit R, De Bono J, Cruz FM, Fountzilas G, Ulys A, Carcano F, Agarwal N, Agus D, Bellmunt J, Petrylak DP, Lee SY, Webb IJ, Tejura B, Borgstein N, Dreicer R. Phase III, randomized, double-blind, multicenter trial comparing orteronel (TAK-700) plus prednisone with placebo plus prednisone in patients with metastatic castration-resistant prostate cancer that has progressed during or after docetaxel-based therapy: ELM-PC 5. J Clin Oncol. 2015 Mar 1;33(7):723-31. doi: 10.1200/JCO.2014.56.5119. Epub 2015 Jan 26. PMID 25624429

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 260 investigative sites in North America, Europe, Argentina, Australia, Brazil, Chile, China, Colombia, Israel, Japan, Mexico, New Zealand, Singapore, South Africa, South Korea, and Taiwan from 15 November 2010 to 29 February 2016.
Pre-assignment Details: Male participants with a historical diagnosis of metastatic-castration resistant prostate cancer (mCRPC) that has progressed during or following docetaxel-based therapy were enrolled in 1 of 2 treatment groups: Orteronel 400 mg + Prednisone 5 mg or Placebo + Prednisone 5 mg.
Groups:
- Placebo + Prednisone: Orteronel placebo-matching tablets, orally, twice daily (BID) and prednisone 5 mg, tablets, orally, BID up to Day 28 of each treatment cycle throughout the study.
- Orteronel + Prednisone: Orteronel 400 mg, tablets, orally, BID and prednisone 5 mg, tablets, orally, BID up to Day 28 of each treatment cycle throughout the study. In Japan only, participants were administered with orteronel 300 mg, tablets, orally, BID and prednisone 5 mg, tablets, orally, BID up to Day 28 of each treatment cycle throughout the study.
Period: Overall Study
Arm/Group | Placebo + Prednisone | Orteronel + Prednisone
Started | 365 | 734
Treated | 363 | 732
Completed | 0 | 0
Not Completed | 365 | 734
Not completed — Death | 202 | 391
Not completed — Study termination by sponsor | 0 | 3
Not completed — Withdrawal by Subject | 26 | 86
Not completed — Lost to Follow-up | 2 | 3
Not completed — Unblinded due to futility | 135 | 251

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all subjects who were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo + Prednisone | Orteronel + Prednisone | Total
Number analyzed (Participants) | 365 | 734 | 1099
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.4 (7.95) | 69.2 (7.82) | 69.3 (7.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 365 | 734 | 1099
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 45 | 107 | 152
  Not Hispanic or Latino | 302 | 588 | 890
  Unknown or Not Reported | 18 | 39 | 57
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 1 | 4 | 5
  Asian | 48 | 77 | 125
  Black or African American | 9 | 18 | 27
  White | 305 | 620 | 925
  Unknown or Not Reported | 1 | 3 | 4
  Other | 1 | 12 | 13
Region of Enrollment [Number; unit: participants]
  Canada | 11 | 21 | 32
  United States | 26 | 54 | 80
  Austria | 5 | 14 | 19
  Belarus | 6 | 4 | 10
  Belgium | 1 | 12 | 13
  Bulgaria | 1 | 3 | 4
  Estonia | 3 | 2 | 5
  Finland | 4 | 7 | 11
  France | 35 | 44 | 79
  Germany | 11 | 35 | 46
  Greece | 22 | 38 | 60
  Hungary | 2 | 7 | 9
  Ireland | 3 | 6 | 9
  Italy | 7 | 14 | 21
  Portugal | 8 | 8 | 16
  Romania | 0 | 12 | 12
  Croatia | 0 | 3 | 3
  Czech Republic | 1 | 1 | 2
  Lithuania | 9 | 22 | 31
  Netherlands | 6 | 12 | 18
  Poland | 5 | 17 | 22
  Russia | 2 | 2 | 4
  Serbia | 1 | 3 | 4
  Slovakia | 5 | 10 | 15
  Spain | 16 | 25 | 41
  Sweden | 10 | 16 | 26
  Switzerland | 1 | 2 | 3
  United Kingdom | 32 | 75 | 107
  Argentina | 1 | 8 | 9
  Australia | 28 | 66 | 94
  Brazil | 37 | 82 | 119
  Chile | 5 | 7 | 12
  China | 5 | 6 | 11
  Colombia | 0 | 4 | 4
  Israel | 5 | 9 | 14
  Japan | 17 | 33 | 50
  Mexico | 1 | 4 | 5
  New Zealand | 6 | 6 | 12
  Singapore | 1 | 1 | 2
  South Africa | 4 | 14 | 18
  Taiwan, Province Of China | 7 | 7 | 14
  Korea, Republic Of | 15 | 18 | 33
Height [Mean (Standard Deviation); unit: centimeter (cm)] — Height data was available for 1096 participants as follows: n= 364, 732.
  centimeter (cm) | 171.33 (7.675) | 172.52 (7.156) | 172.12 (7.350)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] — Weight data was available for 1098 participants as follows: n= 365, 733.
  kilogram (kg) | 79.85 (15.183) | 82.77 (15.200) | 81.80 (15.249)
Body mass index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] — BMI data was available for 1095 participants as follows: n= 364, 731.
  kilogram per square meter (kg/m^2) | 27.14 (4.491) | 27.73 (4.370) | 27.54 (4.418)

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival was calculated from the date of participant randomization to the date of participant death due to any cause. Participants without documentation of death at time of the analysis were censored as of the date the participant was last known to be alive, or the data cutoff date, whichever was earlier.
Time Frame: Baseline until death (approximately up to 4.5 years)
Population: ITT population included all participants who were randomized.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Prednisone | Orteronel + Prednisone
Number analyzed (Participants) | 365 | 734
months | 15.3 [13.48 to 16.86] | 17.1 [15.45 to 18.67]
Statistical Analysis 1: Comparison: Placebo + Prednisone vs Orteronel + Prednisone; Hazard ratio is based on a stratified Cox's proportional hazard regression model with stratification factors region (North America, Europe and Rest of World) and brief pain inventory-short form (BPI-SF) worst pain score at screening ([less than or equal to] <=4, greater than [>] 4) with treatment as a factor in the model. A hazard ratio less than 1 for the treatment indicates better prevention of the death in the Orteronel arm as compared to placebo arm; Test type: Superiority or Other; p = 0.12085, Log Rank; Hazard Ratio (HR) = 0.875, 95% CI 2-sided [0.739 to 1.036]

2. Secondary Outcome: Radiographic Progression-free Survival (rPFS)
Description: rPFS was defined as the time from randomization until radiographic disease progression or death due to any cause, whichever occurred first. Radiographic disease progression was defined as the occurrence of 1 or more of the following: The appearance of 2 or more new lesions on radionuclide bone scan as defined by prostate cancer working group (PCWG)2; Should 2 or more new bone lesions be evident at the first assessment (8-week assessment) on treatment, 2 or more additional new lesions must have been evident on a confirmatory assessment at least 6 weeks later; One or more new soft tissue/visceral organ lesions identified by computed tomography (CT)/magnetic resonance imaging (MRI); Progression as defined by response evaluation criteria in solid tumors (RECIST) 1.1 criteria.
Time Frame: Baseline until disease progression or death, whichever occurred first (approximately up to 4.5 years)
Population: ITT population included all participants who were randomized.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Prednisone | Orteronel + Prednisone
Number analyzed (Participants) | 365 | 734
months | 5.7 [5.46 to 6.97] | 8.3 [7.76 to 8.48]
Statistical Analysis 1: Comparison: Placebo + Prednisone vs Orteronel + Prednisone; Hazard ratio is based on a stratified Cox's proportional hazard regression model with stratification factors region (North America, Europe and Rest of World) and brief pain inventory-short form (BPI-SF) worst pain score at screening (<=4, >4) with treatment as a factor in the model. A hazard ratio less than 1 for the treatment indicates better prevention of the death in the Orteronel arm as compared to placebo arm; Test type: Superiority or Other; p = 0.00038, Log Rank; Hazard Ratio (HR) = 0.760, 95% CI 2-sided [0.653 to 0.885]

3. Secondary Outcome: Percentage of Participants Achieving 50 Percent Reduction From Baseline in Prostate Specific Antigen (PSA50 Response) at Week 12
Description: The PSA50 was defined as the percentage of participants who had a PSA decline of at least 50 percent (%) from baseline.
Time Frame: Week 12
Population: ITT population included all participants who were randomized.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + Prednisone | Orteronel + Prednisone
Number analyzed (Participants) | 365 | 734
percentage of participants | 9.9 | 24.9
Statistical Analysis 1: Comparison: Placebo + Prednisone vs Orteronel + Prednisone; P-values test for odds ratio equal to 1; Test type: Superiority or Other; p < 0.0001, Regression, Logistic

4. Secondary Outcome: Percentage of Participants With Pain Response at Week 12
Description: Pain response was defined as the occurrence of 1 of the following and confirmed by an additional assessment, at least 3 weeks but not more than 5 weeks later: A greater than or equal to (>=) 2 point reduction from baseline in BPI-SF worst pain score without an increase in analgesic use; or a 25 percent (%) or more reduction in analgesic use from baseline without an increase in worst pain score from baseline.
Time Frame: Week 12
Population: ITT population included all participants who were randomized.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + Prednisone | Orteronel + Prednisone
Number analyzed (Participants) | 365 | 734
percentage of participants | 9.0 | 12.1
Statistical Analysis 1: Comparison: Placebo + Prednisone vs Orteronel + Prednisone; P-values test for odds ratio equal to 1; Test type: Superiority or Other; p = 0.12778, Regression, Logistic

5. Secondary Outcome: Number of Participants Reporting One or More Treatment-emergent Adverse Events (TEAEs)
Time Frame: Baseline up to 30 days after last dose of study drug (Cycle 59 Day 58)
Population: Safety population included all participants who received at least 1 dose of any study drug.
Measure: Number; unit: participants
Arm/Group | Placebo + Prednisone | Orteronel + Prednisone
Number analyzed (Participants) | 363 | 732
participants | 345 | 719

6. Secondary Outcome: Number of Participants With Abnormal Physical Examination Findings
Time Frame: Baseline up to 30 days after last dose of study drug (Cycle 59 Day 58)
Population: Safety population included all participants who received at least 1 dose of any study drug.
Measure: Number; unit: participants
Arm/Group | Placebo + Prednisone | Orteronel + Prednisone
Number analyzed (Participants) | 363 | 732
participants | 0 | 1

7. Secondary Outcome: Number of Participants With TEAEs Related to Vital Signs
Time Frame: Baseline up to 30 days after last dose of study drug (Cycle 59 Day 58)
Population: Safety population included all participants who received at least 1 dose of any study drug.
Measure: Number; unit: participants
Arm/Group | Placebo + Prednisone | Orteronel + Prednisone
Number analyzed (Participants) | 363 | 732
participants
  Hypertension | 21 | 83
  Hypotension | 8 | 31
  Pyrexia | 18 | 51

8. Secondary Outcome: Number of Participants With TEAEs Related to Weight
Time Frame: Baseline up to 30 days after last dose of study drug (Cycle 59 Day 58)
Population: Safety population included all participants who received at least 1 dose of any study drug.
Measure: Number; unit: participants
Arm/Group | Placebo + Prednisone | Orteronel + Prednisone
Number analyzed (Participants) | 363 | 732
participants
  Weight decreased | 32 | 107
  Weight increased | 7 | 6

9. Secondary Outcome: Number of Participants With Worst Change From Baseline in Eastern Co-operative Oncology Group (ECOG) Performance Status
Description: ECOG assessed participant's performance status on 5 point scale: 0=Fully active/able to carry on all pre-disease activities without restriction; 1=restricted in physically strenuous activity, ambulatory/able to carry out light or sedentary work; 2=ambulatory (>50% of waking hours [hrs]), capable of all self care, unable to carry out any work activities; 3=capable of only limited self care, confined to bed/chair >50% of waking hrs; 4=completely disabled, cannot carry on any self care, totally confined to bed/chair; 5=dead. Worst change was defined as the worst overall change that occurred in ECOG status at any measured time point during the treatment period.
Time Frame: Baseline up to End-of-treatment (EOT) (Cycle 59 Day 58)
Population: Safety population where baseline and post-baseline assessments were available. Safety population included all participants who received at least 1 dose of any study drug.
Measure: Number; unit: participants
Arm/Group | Placebo + Prednisone | Orteronel + Prednisone
Number analyzed (Participants) | 353 | 705
participants
  Baseline: 0; Overall: 0 | 56 | 112
  Baseline: 0; Overall: 1 | 70 | 121
  Baseline: 0; Overall: 2 | 13 | 47
  Baseline: 0; Overall: 3 | 5 | 18
  Baseline: 0; Overall: 4 | 1 | 3
  Baseline: 1; Overall: 0 | 3 | 10
  Baseline: 1; Overall: 1 | 103 | 179
  Baseline: 1; Overall: 2 | 53 | 113
  Baseline: 1; Overall: 3 | 22 | 39
  Baseline: 1; Overall: 4 | 7 | 11
  Baseline: 2; Overall: 1 | 0 | 6
  Baseline: 2; Overall: 2 | 10 | 25
  Baseline: 2; Overall: 3 | 10 | 18
  Baseline: 2; Overall: 4 | 0 | 3

10. Secondary Outcome: Number of Participants With Abnormal Clinically Significant Electrocardiogram (ECG) Findings
Time Frame: Cycle 59 Day 58
Population: Safety population included all participants who received at least 1 dose of any study drug.
Measure: Number; unit: participants
Arm/Group | Placebo + Prednisone | Orteronel + Prednisone
Number analyzed (Participants) | 363 | 732
participants | 1 | 3

11. Secondary Outcome: Number of Participants With TEAEs Categorized Into Investigations Related to Chemistry, Hematology or Steroid Hormone Panel
Time Frame: Baseline up to 30 days after last dose of study drug (Cycle 59 Day 58)
Population: Safety population included all participants who received at least 1 dose of any study drug.
Measure: Number; unit: participants
Arm/Group | Placebo + Prednisone | Orteronel + Prednisone
Number analyzed (Participants) | 363 | 732
participants
  Digestive enzymes | 9 | 140
  Renal function analyses | 13 | 41
  Liver function analyses | 14 | 38
  Tissue enzyme analyses NEC | 16 | 30
  Coagulation and bleeding analyses | 1 | 17
  Mineral and electrolyte analyses | 5 | 9
  White blood cell analyses | 4 | 8
  Carbohydrate tolerance analyses-including diabetes | 0 | 8
  Urinary tract function analyses NEC | 1 | 5
  Platelet analyses | 3 | 4
  Cholesterol analyses | 1 | 4
  Red blood cell analyses | 2 | 3
  Protein analyses not elsewhere classified (NEC) | 0 | 3
  Vascular tests NEC (including blood pressure) | 3 | 2
  Adrenal cortex tests | 0 | 2
  Metabolism tests NEC | 0 | 2
  Skeletal and cardiac muscle analyses | 0 | 2
  Triglyceride analyses | 0 | 1
  Urinalysis NEC | 0 | 1
  Vitamin analyses | 0 | 1

12. Secondary Outcome: Percentage of Participants Achieving PSA50 Response at Any Time During the Study
Description: The PSA50 was defined as the percentage of participants who had a PSA decline of at least 50% from baseline.
Time Frame: Cycle: 4, 7, 10, 13, 16, 19, 22, and 25
Population: ITT population where baseline and post-baseline assessments were available. The ITT population included all participants who were randomized.
Measure: Number; unit: participants
Arm/Group | Placebo + Prednisone | Orteronel + Prednisone
Number analyzed (Participants) | 365 | 734
participants
  Cycle 4 (n= 283; 559) | 12.72 | 32.74
  Cycle 7 (n= 163; 403) | 18.40 | 38.21
  Cycle 10 (n= 102; 267) | 22.55 | 36.70
  Cycle 13 (n= 55; 171) | 23.64 | 40.94
  Cycle 16 (n= 34; 107) | 23.53 | 44.86
  Cycle 19 (n= 24; 68) | 20.83 | 42.65
  Cycle 22 (n= 14; 36) | 28.57 | 52.78
  Cycle 25 (n= 8; 16) | 25.00 | 62.50

13. Secondary Outcome: Percentage of Participants Achieving 90 Percent Reduction From Baseline in Prostate Specific Antigen (PSA90 Response) at Week 12
Description: The PSA90 was defined as the percentage of participants who had a PSA decline of at least 90% from baseline.
Time Frame: Week 12
Population: ITT population where baseline and post-baseline assessments were available. ITT population included all participants who were randomized.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + Prednisone | Orteronel + Prednisone
Number analyzed (Participants) | 283 | 559
percentage of participants | 2.83 | 9.66

14. Secondary Outcome: Percentage of Participants Achieving PSA90 Response at Any Time During the Study
Description: The PSA90 was defined as the percentage of participants who had a PSA decline of at least 90% from baseline.
Time Frame: Cycle: 7, 10, 13, 16, 19, 22, and 25
Population: as for outcome 13
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + Prednisone | Orteronel + Prednisone
Number analyzed (Participants) | 365 | 734
percentage of participants
  Cycle 7 (n=163; 403) | 4.91 | 14.89
  Cycle 10 (n=102; 267) | 6.86 | 14.23
  Cycle 13 (n=55; 171) | 7.27 | 15.20
  Cycle 16 (n=34; 107) | 5.88 | 19.63
  Cycle 19 (n=24; 68) | 4.17 | 23.53
  Cycle 22 (n=14; 36) | 0.00 | 27.78
  Cycle 25 (n=8; 16) | 0.00 | 43.75

15. Secondary Outcome: Best PSA Response at Any Time During the Study
Description: The PSA50 was defined as the percentage of participants who had a PSA decline of at least 50% from baseline. PSA90 was defined as the percentage of participants who had a PSA decline of at least 90% from baseline.
Time Frame: Cycle: 4, 7, 10, 13, 16, 19, 22, and 25
Population: Best PSA response was not evaluated due to change in planned analysis.
Arm/Group | Placebo + Prednisone | Orteronel + Prednisone
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Time to PSA Progression
Description: Time to PSA progression was defined as time from randomization to a PSA increase of 25% and PSA rise of at least 2 nanogram per milliliter (ng/mL) above the lowest value observed post baseline or, if no PSA decline occurred post baseline, above the baseline PSA.
Time Frame: Baseline until the final on treatment assessment or until end of short term follow-up following discontinuation of treatment, whichever occurred later (approximately up to 4.5 years)
Population: ITT population included all participants who were randomized.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Prednisone | Orteronel + Prednisone
Number analyzed (Participants) | 365 | 734
months | 2.9 [2.83 to 2.90] | 5.5 [4.40 to 5.56]

17. Secondary Outcome: Number of Participants With Shifts From Baseline Between Favorable and Unfavorable Categories in Circulating Tumor Cell Count (CTC)
Description: A favorable CTC count was defined as less than (<) 5 counts per (/) 7.5 mililiter (mL) in whole blood. An unfavorable CTC count was defined as >=5 counts/7.5 mL in whole blood.
Time Frame: Baseline and EOT (Cycle 59 Day 58)
Population: as for outcome 13
Measure: Number; unit: participants
Arm/Group | Placebo + Prednisone | Orteronel + Prednisone
Number analyzed (Participants) | 157 | 267
participants
  Baseline: Favorable; EOT: Favorable | 27 | 63
  Baseline: Favorable; EOT: Unfavorable | 30 | 40
  Baseline: Unfavorable; EOT: Favorable | 8 | 23
  Baseline: Unfavorable; EOT: Unfavorable | 92 | 141

18. Secondary Outcome: Percentage of Participants With Objective Response
Description: Percentage of participants with objective response based assessment of confirmed complete response (CR) or confirmed partial response (PR) according to RECIST 1.1. The overall objective response was defined as a complete response (CR) or partial response (PR). A complete response (CR) was defined as the disappearance of all target lesions determined by computerized tomography (CT) or MRI. Any pathological lymph nodes (whether target or non-target) must have had reduction in short axis to <10 millimetre (mm). A PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of longest diameters of non-lymph node lesions and of the short diameter(s) or short axis of lymph nodes.
Time Frame: Baseline until disease progression or death, whichever occurred first (approximately up to 4.5 years)
Population: Response per RECIST-evaluable population was defined as a subset of participants who had measurable disease by RECIST 1.1 at baseline.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + Prednisone | Orteronel + Prednisone
Number analyzed (Participants) | 146 | 280
percentage of participants | 2.7 | 17.1

19. Secondary Outcome: Time to Pain Progression
Description: Time to pain progression was defined as the time from participant randomization to the first assessment date of pain progression. Pain progression was defined as the occurrence of 1 of the following and confirmed by an additional assessment, at least 3 weeks but not more than 5 weeks later: The brief pain inventory-short form (BPI-SF) worst pain score was >= 4 with a >= 2 point increase over baseline in BPI-SF worst pain score with stable or increased analgesic use; The BPI-SF worst pain score was >= 4 but not less than baseline with new or increased (relative to baseline) Step II or Step III analgesic use; The BPI-SF worst pain score was <= 3 but not less than baseline with new or increased (relative to baseline) Step III analgesic use.
Time Frame: Baseline until EOT visit or until end of short term follow-up, whichever occurred later (approximately up to 4.5 years)
Population: ITT population included all participants who were randomized.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Prednisone | Orteronel + Prednisone
Number analyzed (Participants) | 365 | 734
months | 22.0 [20.48 to NA] — The upper limit was not estimable. | 24.2 [18.24 to 24.20]

20. Secondary Outcome: Time to Pain Response
Description: Time to pain response was defined as the time from randomization until first pain response. Pain response was defined as the occurrence of 1 of the following and confirmed by an additional assessment, at least 3 weeks but not more than 5 weeks later: A >= 2 point reduction from baseline in BPI-SF worst pain score without an increase in analgesic use, or a 25% or more reduction in analgesic use from baseline without an increase in worst pain score from baseline. The analysis was performed by Kaplan-Meier method.
Time Frame: Baseline until disease progression or death, whichever occurred first (approximately up to 4.5 years)
Population: ITT population included all participants who were randomized.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Prednisone | Orteronel + Prednisone
Number analyzed (Participants) | 365 | 734
months | NA [NA to NA] — Median: No data is reported since median time to pain response was not estimable (that is, not reached) in either treatment group due to low number of events. Confidence interval: Confidence interval was not estimable due to low number of events | NA [NA to NA] — Median: No data is reported since median time to pain response was not estimable (that is, not reached) in either treatment group due to low number of events. Confidence interval: Confidence interval was not estimable due to low number of events

21. Secondary Outcome: Number of Participants With Best Pain Response
Description: Best pain response was evaluated in participants who had a pain response across the entire study were summarized by treatment group. The pain response was defined as a >=2-point reduction from baseline in BPI-SF worst pain score without an increase in analgesic use, or a 25% or more reduction in analgesic use from baseline without an increase in worst pain score from baseline.
Time Frame: Baseline until disease progression or death, whichever occurred first (approximately up to 4.5 years)
Population: ITT population included all participants who were randomized.
Measure: Number; unit: participants
Arm/Group | Placebo + Prednisone | Orteronel + Prednisone
Number analyzed (Participants) | 365 | 734
participants | 72 | 166

22. Secondary Outcome: Percentage of Participants With Health-related Quality of Life (HRQOL) Response at Week 12
Description: The global health status or quality of life (QOL) was measured as the HRQOL response rate at 12 weeks using the 2-item global health status index of the european organization for research and treatment of cancer-quality of life questionnaire-C30 (EORTC QLQ-C30) instrument. HRQOL response was defined as a 17-point increase from the baseline assessment on the QOL index, after the score had been linearly transformed to a 0 to 100 scale. EORTC QLQ-C30: included 5 functional scales (physical, role, cognitive, emotional, and social), 1 global health status, 3 symptom scales (fatigue, pain, nausea/vomiting) and 6 single items (dyspnoea, appetite loss, insomnia, constipation/diarrhea and financial difficulties). Most questions used 4 point scale (1 'Not at all' to 4 'Very much'; 2 questions used 7-point scale (1 'very poor' to 7 'Excellent'). Scores averaged, transformed to 0-100 scale; higher score representing better level of functioning or greater degree of symptoms.
Time Frame: Week 12
Population: ITT population included all participants who were randomized.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + Prednisone | Orteronel + Prednisone
Number analyzed (Participants) | 365 | 734
percentage of participants | 9.9 | 8.7

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of double-blind study drug and no more than 30 days (Cycle 59 Day 58) after the last dose of study drug.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Placebo + Prednisone | Orteronel + Prednisone
Serious Adverse Events (participants affected / at risk) | 148/363 | 384/732
Other Adverse Events (participants affected / at risk) | 341/363 | 703/732
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + Prednisone (N=363) | Orteronel + Prednisone (N=732)
Sepsis (Infections and infestations) | 3 | 14
Urosepsis (Infections and infestations) | 2 | 12
Septic shock (Infections and infestations) | 4 | 7
Bacteraemia (Infections and infestations) | 0 | 3
Pneumonia (Infections and infestations) | 9 | 19
Lower respiratory tract infection (Infections and infestations) | 2 | 3
Lung infection (Infections and infestations) | 1 | 3
Bronchopneumonia (Infections and infestations) | 0 | 3
Lobar pneumonia (Infections and infestations) | 0 | 3
Urinary tract infection (Infections and infestations) | 4 | 20
Pyelonephritis (Infections and infestations) | 0 | 4
Pyelonephritis acute (Infections and infestations) | 0 | 1
Pyelonephritis chronic (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 3
Gastroenteritis (Infections and infestations) | 1 | 2
Anal abscess (Infections and infestations) | 0 | 2
Abdominal infection (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Peritonitis (Infections and infestations) | 0 | 1
Rectal abscess (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 5
Pneumonia bacterial (Infections and infestations) | 1 | 1
Bacterial infection (Infections and infestations) | 0 | 1
Endocarditis bacterial (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 1 | 1
Respiratory tract infection (Infections and infestations) | 1 | 1
Infection (Infections and infestations) | 0 | 1
Pelvic abscess (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 3
Staphylococcal bacteraemia (Infections and infestations) | 1 | 2
Staphylococcal sepsis (Infections and infestations) | 1 | 0
Abscess oral (Infections and infestations) | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 1
Escherichia bacteraemia (Infections and infestations) | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 0 | 1
Soft tissue infection (Infections and infestations) | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 0 | 1
Pneumonia pneumococcal (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Fungal oesophagitis (Infections and infestations) | 0 | 1
Proteus infection (Infections and infestations) | 0 | 1
Salmonella sepsis (Infections and infestations) | 0 | 1
Spinal cord infection (Infections and infestations) | 1 | 0
Nosocomial infection (Infections and infestations) | 1 | 0
Listeriosis (Infections and infestations) | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 24 | 33
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 6
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 9
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 5
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Metastatic pulmonary embolism (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to the mediastinum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bone marrow tumour cell infiltration (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Anal cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Vomiting (Gastrointestinal disorders) | 6 | 18
Nausea (Gastrointestinal disorders) | 0 | 13
Abdominal pain (Gastrointestinal disorders) | 3 | 10
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 3 | 6
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 3
Pancreatitis acute (Gastrointestinal disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 5
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 3
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Subileus (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 2
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 2
Gastroduodenitis (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 3
Haematochezia (Gastrointestinal disorders) | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Oesophageal haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Ileus paralytic (Gastrointestinal disorders) | 0 | 1
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastritis erosive (Gastrointestinal disorders) | 1 | 0
Diverticulitis intestinal haemorrhagic (Gastrointestinal disorders) | 1 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 1 | 0
General physical health deterioration (General disorders) | 4 | 19
Multi-organ failure (General disorders) | 0 | 3
Disease progression (General disorders) | 0 | 2
Performance status decreased (General disorders) | 0 | 1
Fatigue (General disorders) | 4 | 10
Asthenia (General disorders) | 3 | 10
Malaise (General disorders) | 1 | 4
Pyrexia (General disorders) | 2 | 8
Pain (General disorders) | 2 | 3
Chest pain (General disorders) | 1 | 2
Non-cardiac chest pain (General disorders) | 0 | 2
Spinal pain (General disorders) | 0 | 0
Oedema peripheral (General disorders) | 0 | 3
Generalised oedema (General disorders) | 0 | 1
Death (General disorders) | 0 | 1
Sudden death (General disorders) | 1 | 0
Thrombosis in device (General disorders) | 1 | 1
Device occlusion (General disorders) | 0 | 1
Systemic inflammatory response syndrome (General disorders) | 0 | 1
Drug intolerance (General disorders) | 0 | 1
Gait disturbance (General disorders) | 1 | 0
Cyst (General disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 4 | 12
Renal failure (Renal and urinary disorders) | 0 | 11
Postrenal failure (Renal and urinary disorders) | 0 | 3
Renal impairment (Renal and urinary disorders) | 2 | 2
Chronic kidney disease (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 3 | 14
Dysuria (Renal and urinary disorders) | 0 | 2
Urge incontinence (Renal and urinary disorders) | 0 | 1
Micturition urgency (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 3 | 9
Hydronephrosis (Renal and urinary disorders) | 3 | 3
Obstructive uropathy (Renal and urinary disorders) | 1 | 0
Renal disorder (Renal and urinary disorders) | 1 | 2
Azotaemia (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Calculus urethral (Renal and urinary disorders) | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 4 | 0
Urinoma (Renal and urinary disorders) | 1 | 0
Bladder perforation (Renal and urinary disorders) | 1 | 0
Ureteric rupture (Renal and urinary disorders) | 1 | 0
Spinal cord compression (Nervous system disorders) | 9 | 17
Cauda equina syndrome (Nervous system disorders) | 1 | 0
Nerve root compression (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 2 | 8
Lethargy (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 5
Presyncope (Nervous system disorders) | 1 | 4
Paraparesis (Nervous system disorders) | 1 | 4
Paraplegia (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 1
Cerebral ischaemia (Nervous system disorders) | 0 | 1
Haemorrhagic stroke (Nervous system disorders) | 0 | 1
Intraventricular haemorrhage (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1
Central nervous system haemorrhage (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Vascular encephalopathy (Nervous system disorders) | 0 | 1
Vertebrobasilar insufficiency (Nervous system disorders) | 0 | 1
Ataxia (Nervous system disorders) | 0 | 1
Hepatic encephalopathy (Nervous system disorders) | 0 | 1
VIIth nerve paralysis (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 1
Parkinson's disease (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 1 | 0
Neuralgia (Nervous system disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 20
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 8
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 7
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alveolitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 10
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1
Flank pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 14 | 8
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Pubic pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 7
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 4
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 3
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 | 3
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 | 2
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 2
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 2 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 5
Myocardial infarction (Cardiac disorders) | 2 | 4
Angina unstable (Cardiac disorders) | 0 | 2
Myocardial ischaemia (Cardiac disorders) | 0 | 2
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 9
Atrial flutter (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 5
Cardiopulmonary failure (Cardiac disorders) | 1 | 1
Cardiac failure acute (Cardiac disorders) | 0 | 1
Cardiac failure chronic (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 4
Cardiac arrest (Cardiac disorders) | 1 | 3
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 2
Left ventricular dysfunction (Cardiac disorders) | 1 | 1
Aortic valve stenosis (Cardiac disorders) | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 15
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 10
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 10
Decreased appetite (Metabolism and nutrition disorders) | 4 | 4
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 2
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 2
Cachexia (Metabolism and nutrition disorders) | 0 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 9 | 21
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 3
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 2
Anaemia of chronic disease (Blood and lymphatic system disorders) | 0 | 1
Anaemia of malignant disease (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 1
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 0 | 1
Lipase increased (Investigations) | 1 | 12
Amylase increased (Investigations) | 1 | 5
Pancreatic enzymes increased (Investigations) | 0 | 4
Liver function test abnormal (Investigations) | 0 | 3
Alanine aminotransferase increased (Investigations) | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 1 | 2
International normalised ratio increased (Investigations) | 0 | 2
Blood cortisol decreased (Investigations) | 0 | 1
Blood glucose increased (Investigations) | 0 | 1
Weight decreased (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 3
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 3
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 3
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Radiation proctitis (Injury, poisoning and procedural complications) | 0 | 1
Transfusion-related circulatory overload (Injury, poisoning and procedural complications) | 0 | 1
Kidney rupture (Injury, poisoning and procedural complications) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0
Hypotension (Vascular disorders) | 0 | 3
Orthostatic hypotension (Injury, poisoning and procedural complications) | 0 | 1
Deep vein thrombosis (Injury, poisoning and procedural complications) | 3 | 3
Haemorrhage (Vascular disorders) | 0 | 2
Embolism (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 2
Hypertensive crisis (Vascular disorders) | 0 | 1
Lymphoedema (Vascular disorders) | 0 | 1
Phlebitis (Vascular disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 4
Depression (Psychiatric disorders) | 0 | 2
Delusion (Psychiatric disorders) | 0 | 1
Psychotic disorder (Psychiatric disorders) | 0 | 1
Delirium (Psychiatric disorders) | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 3
Mineralocorticoid deficiency (Endocrine disorders) | 0 | 1
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 3
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 0 | 1
Cholestasis (Hepatobiliary disorders) | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Bile duct stenosis (Hepatobiliary disorders) | 1 | 0
Prostatomegaly (Reproductive system and breast disorders) | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 1
Diplopia (Eye disorders) | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Cor pulmonale (Cardiac disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + Prednisone (N=363) | Orteronel + Prednisone (N=732)
Anaemia (Blood and lymphatic system disorders) | 59 | 103
Nausea (Gastrointestinal disorders) | 94 | 319
Vomiting (Gastrointestinal disorders) | 60 | 272
Constipation (Gastrointestinal disorders) | 64 | 222
Diarrhoea (Gastrointestinal disorders) | 54 | 201
Abdominal pain (Gastrointestinal disorders) | 21 | 46
Dyspepsia (Gastrointestinal disorders) | 13 | 46
Fatigue (General disorders) | 84 | 223
Asthenia (General disorders) | 39 | 102
Oedema peripheral (General disorders) | 45 | 77
Pyrexia (General disorders) | 18 | 48
Urinary tract infection (Infections and infestations) | 24 | 57
Weight decreased (Investigations) | 34 | 113
Lipase increased (Investigations) | 5 | 113
Amylase increased (Investigations) | 5 | 101
Blood creatinine increased (Investigations) | 9 | 38
Decreased appetite (Metabolism and nutrition disorders) | 68 | 208
Hypokalaemia (Metabolism and nutrition disorders) | 14 | 45
Back pain (Musculoskeletal and connective tissue disorders) | 62 | 139
Arthralgia (Musculoskeletal and connective tissue disorders) | 55 | 112
Bone pain (Musculoskeletal and connective tissue disorders) | 51 | 89
Muscle spasms (Musculoskeletal and connective tissue disorders) | 27 | 110
Pain in extremity (Musculoskeletal and connective tissue disorders) | 45 | 86
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 24 | 57
Myalgia (Musculoskeletal and connective tissue disorders) | 20 | 39
Muscular weakness (Musculoskeletal and connective tissue disorders) | 21 | 36
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 16 | 39
Headache (Nervous system disorders) | 23 | 76
Dizziness (Nervous system disorders) | 15 | 78
Insomnia (Psychiatric disorders) | 26 | 67
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 21 | 67
Cough (Respiratory, thoracic and mediastinal disorders) | 19 | 63
Hypertension (Vascular disorders) | 22 | 84
Hot flush (Vascular disorders) | 20 | 63

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In general, Investigators may publish clinical data after the earlier of (i) publication by the Sponsor or (ii) 12 months following the abandonment, early termination or database lock; provided a copy of the publication provided to Sponsor at least 30 days ahead of publication, the Sponsor's confidential information is removed as may be requested by Sponsor and Investigator defers publication for up to 60 days in the event Sponsor provides notice that it intends to file a patent application.